CLINICAL TRIAL: NCT04511442
Title: Comparative Study of Differences in Food Preferences and Sensory Perceptions Between People With Obesity With or Without Bariatric Surgery
Brief Title: Study of Food Preferences and Sensory Perceptions After Bariatric Surgery
Acronym: BariaTaste 2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0182
Record Dates: First submitted 2020-07-16; First posted 2020-08-13 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric surgery: Women with obesity, with a bariatric surgery
  Interventions: Other: Evaluation of food preferences during a standardized and validated buffet.
- Control: Women with obesity, without a bariatric surgery
  Interventions: Other: Evaluation of food preferences during a standardized and validated buffet.

INTERVENTIONS:
Other: Evaluation of food preferences during a standardized and validated buffet. — The dietary preferences of people will be collected by a direct measurement of eating behavior in front of a dedicated and standardized ad-libitum buffet.
  As part of this buffet, 3 dichotomous categories of food will be studied:
  * high / low in fat (HF / LF)
  * high / low in carbohydrates (HC / LC)
  * high / low in protein (HP / LP). During the buffet, participants will be filmed to study their food choices and the microstructure of their meal. We will define food preferences as the relative consumption choices of the food categories studied. We will also collect the time spent at the buffet, the duration of ingestion, the total duration of the meal, the number of bites per minute, the total number of bites and the number of bites by type of food.
  Weighing's will be carried out before and after consumption in order to determine the total energy intake and the macronutrient intake (proteins, lipids, carbohydrates) of the participants.

SUMMARY:
Several studies report changes in food preferences in favor of low energy density foods after bariatric surgery and changes in scores of liking and desire to eat, as well as changes in hedonic evaluation certain foods. However, only one study was held in a more realistic condition of consumption by using real food, looking at some aspects of food preferences and giving contradictory results. We hypothesise that food preferences are different between obese people with and without a bariatric surgery. The main objective of this study is to compare the differences in food quality (proportion of total energy intake from foods with high energy density versus foods with low energy density), evaluated during a standardized and validated buffet between adult women with severe complicated or morbid obesity and women who have undergone bariatric surgery in the last 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Woman from 18 to 65 years old (included)
* Person capable of going to the Institut Paul Bocuse Research Center, Bellecour platform, 20 Place Bellecour, 69002 Lyon
* Person who agree to participate in the study
* Person having signed the consent of image rights
* For the surgery group: person who has undergone bariatric surgery (except gastric band)
* For the control group: person with a BMI ≥ 35 kg / m2 who did not benefit from bariatric surgery

Exclusion Criteria:

* Person with a food allergy or food intolerance to at least one of the study products
* Person excluding certain foods from their diet for religious or personal reasons.
* Person who smoke
* Person with severe digestive disorders, dysphagia, abdominal pain
* Person who cannot give her agreement, not mastering the French language
* Person who has exceeded the annual amount of compensation in the year for participation in research protocols
* Pregnant or breastfeeding woman or not taking effective contraception
* Person with a history of pathology which may interfere according to the investigator with the criteria of the study (ENT, neurological, upper digestive pathologies, ...)
* For the surgery group: conversion of any type of bariatric surgery

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: This study will focus on adult female volunteers with severe complicated or morbid obesity who may or may not have undergone bariatric surgery in the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2021-12-21 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Food preference for high energy dense foods | Day 1
  The main endpoint of the study is the proportion of total energy intake from foods with high energy density versus foods with low energy density evaluated during a standardized and validated buffet.

CONTACTS AND LOCATIONS:
Locations (1):
- : Center for Research in Human Nutrition Rhône-Alpes, Institut Paul Bocuse Research Center, Lyon, France